CLINICAL TRIAL: NCT05294406
Title: Evaluation of a Pilot Implementation of Intermittent Preventive Treatment With Dihydroartemisinin-piperaquine to Prevent Adverse Birth Outcomes in Papua, Indonesia
Brief Title: Intermittent Preventive Treatment With Dihydroartemisinin-piperaquine in Papua, Indonesia
Acronym: STOPMiP-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Gadjah Mada University (Other); Indonesia-MoH (Other Government); Yayasan Pengembangan Kesehatan dan Masyarakat Papua (Timika Research Facility) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 21-054
Record Dates: First submitted 2022-03-09; First posted 2022-03-24 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Malaria in Pregnancy
MeSH Terms: interventions — Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IPTp-DP (Experimental): Pregnant women attending routine antenatal care visits in their second and third trimester are given a monthly, presumptive treatment dose of dihydroartemisinin-piperaquine of three tablets daily for three days (9 tablets). The first dose is given by directly observed therapy (DOT), and the remaining doses given to the women to take at home.
  Interventions: Drug: Intermittent preventive treatment in pregnancy (IPTp) with dihydroartemisinin-piperaquine

INTERVENTIONS:
Drug: Intermittent preventive treatment in pregnancy (IPTp) with dihydroartemisinin-piperaquine — Pregnant women attending routine antenatal care visits in their second and third trimester are given monthly IPTp consisting of a treatment dose of dihydroartemisinin-piperaquine (3 tablets per day for 3 days, 9 tablets total)

SUMMARY:
Malaria in pregnancy is a major cause of maternal and neonatal death in Papua, Indonesia. A recent trial in Papua showed that monthly intermittent preventive treatment (IPTp) with the long-acting artemisinin-based combination dihydroartemisinin-piperaquine (DP) among pregnant women in the second and third trimester was safe, tolerable and more efficacious than the current policy of single screening at antenatal care (ANC) booking and treatment of rapid diagnostic test (RDT)-positive cases. The Ministry of Health (MOH) Indonesia now plans to pilot the strategy in the routine health system in Papua, Indonesia. This study will assess the programme effectiveness of IPTp-DP delivery through antenatal care services and women's adherence to the monthly 3-day DP treatment regimen in a 'real life' setting.

The study will be undertaken in ten community health centres in the lowlands and their associated health posts in Timika city. In the first 18 months, MOH will be trained to implement the intervention using quality improvement (QI) approaches to continuously strengthen service delivery, uptake and adherence through plan-do-study-act cycles. The MOH will also be supported to collect safety data for pharmacovigilance. A mixed-methods evaluation will be conducted towards the end of the pilot using exit interviews to assess delivery effectiveness, home visits to assess adherence, and qualitative research to explore provider perceptions of the drivers of successful integration and scalability, and user acceptability. The primary outcome is adherence, defined as the proportion of pregnant women who receive the first dose of IPTp-DP by directly observed therapy (DOT) at ANC, have received the correct number of DP tablets for subsequent doses, and when visited at home have verified they completed the course. The net cost-effectiveness of implementing IPTp-DP and of the current policy of single screening and treatment (SST) in the routine health system will be assessed and compared. Net cost-effectiveness means that cost savings from averted malaria will be deducted from the intervention costs. The incremental financial cost of implementing IPTp-DP from the provider (MOH) perspective at scale in Papua, Indonesia, will also be estimated.

ELIGIBILITY:
Inclusion Criteria:

Health facilities (pilot implementation)

* Antenatal services must be operational and accessible
* Midwives/nurses have been trained to prescribe IPTp-DP

Healthcare providers

* Healthcare providers responsible for providing antenatal care services, and facility managers
* District and provincial health managers

Pregnant women

* Pregnant women aged 15-49 years
* Women in 2nd/3rd trimester of pregnancy
* HIV negative (where status is known)

Community members

* community leaders
* community health care workers
* husbands of pregnant women

Exclusion Criteria:

Health facilities (pilot implementation)

* Health facilities which have accessibility issues and will not be enrolled in the pilot.

Healthcare providers

* Health workers providing ANC and IPTp-DP services in health facilities who have provided services for <1 month.

Pregnant women

* Women with communication or language problems including not being able to speak Indonesian.
* Pregnant women who are unwell during interview
* Pregnant women who move outside the pilot implementation areas.

Ages: 15 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2128 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Adherence in pregnant women | At study completion, an average of 10 months
  The proportion of pregnant women who receive the first dose of IPTp-DP by DOT at ANC clinic and have the correct number of DP tablets for subsequent doses on exiting, who when visited at home verify they have completed the treatment (self report and pill counts)
Delivery effectiveness | At study completion, an average of 10 months
  The proportion of women attending ANC clinic treated appropriately according to the IPTp-DP guidelines, defined as the first dose given by directly observed therapy (DOT) on day-1 plus adequate doses to take home for days 2 and 3. Women's understanding of the treatment regimens given during that ANC visit will also be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Hill, MSc, PhD, Principal Investigator — LSTM
Locations (1):
- Yayasan Pengembangan Kesehatan dan Masyarakat Papua, Timika, Special Region of Papua, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hafidz F, Candrawati F, Hoyt J, Kenangalem E, Dodd J, Lesosky M, Laksanawati IS, Ubra R, Simatupang M, Ter Kuile FO, Worrall E, Poespoprodjo JR, Hill J. Pilot implementation of intermittent preventive treatment with dihydroartemisinin-piperaquine to prevent adverse birth outcomes in Papua, Indonesia: a mixed-method evaluation. Lancet Prim Care. 2025 Jul;1(1):None. doi: 10.1016/j.lanprc.2025.100011. PMID 40874017